CLINICAL TRIAL: NCT02879747
Title: Individualizing the Dose of Growth Hormone (GH) to Maintain Normal Growth Velocity After Fulfilled Catch up Growth in Children Within TR 98-0198-003
Brief Title: Individualizing Dose of Growth Hormone to Maintain Normal Growth Velocity After Fulfilled Catch up Growth in Children
Acronym: MAINTENANCE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRA 6280003
Record Dates: First submitted 2016-08-10; First posted 2016-08-26 (Estimated); Results first posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Short Stature
Keywords: treatment; growth hormone; childhood; short stature
MeSH Terms: conditions — Dwarfism | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interventional (Active Comparator): Unchanged dose Genotropin
  Interventions: Drug: Genotropin
- Interventional 2 (Active Comparator): reduced dose 50% Genotropin
  Interventions: Drug: Genotropin

INTERVENTIONS:
Drug: Genotropin — Children were randomized to either decreased dose by 50% or unchanged dose after 2-3 years of Catch-up growth

SUMMARY:
The objective was to study whether normal growth velocity can be maintained with adapted GH dosage in GH treated prepubertal children who have responded to GH treatment with fulfilled catch up growth (=difference to target height reached, less than - 0.6 SDS).

DETAILED DESCRIPTION:
The aim of the trial is to study the effect of adapted GH treatment in order to find an individualized GH dose maintaining normal growth velocity close to target height SDS and normal metabolism after fulfilled catch up growth in prepubertal children treated with individual doses of GH within the trial 98-0198-003 (1). The overall aim is to find for the individual the lowest effective GH dose during maintenance period, maintaining normal growth velocity and metabolism, i.e. a satisfactory biological active dose.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the 'GH-dose catch-up study' 98- 0198-003.
* Midparental height reached (difference less than 0.6 SDS)
* Prepubertal at start of the study (girls =B 1, boys: testes :<; 3ml).
* Signed written informed consent from the patient's parents (and the child if old enough)

Exclusion Criteria:

* Disease affecting growth other than correctly treated hypothyroidism.
* Incapable of following the study protocol (i.e. bad compliance in the previous study).
* Puberty (> breast stage 2, or testes > 4ml).
* Poor compliance.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 99 (Actual)
Dates: Start 2003-12 (Actual); Primary Completion 2012-03 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Berit Kriström, MD, Principal Investigator — Umeå University Hospital; Nils-Östen Nilsson, MD, Principal Investigator — Halmstad Department of Pediatrics; Maria Halldin, MD, Principal Investigator — Uppsala University Hospital; Sten Ivarsson, MD, Prof, Principal Investigator — Malmö Academic Hospital; Kerstin Albertsson-Wikland, MD, prof, Principal Investigator — Gothenburg University, Departments of pediatrics

REFERENCES:
- [Background] Wikland KA, Kristrom B, Rosberg S, Svensson B, Nierop AF. Validated multivariate models predicting the growth response to GH treatment in individual short children with a broad range in GH secretion capacities. Pediatr Res. 2000 Oct;48(4):475-84. doi: 10.1203/00006450-200010000-00010. PMID 11004238
- [Result] Kristrom B, Aronson AS, Dahlgren J, Gustafsson J, Halldin M, Ivarsson SA, Nilsson NO, Svensson J, Tuvemo T, Albertsson-Wikland K. Growth hormone (GH) dosing during catch-up growth guided by individual responsiveness decreases growth response variability in prepubertal children with GH deficiency or idiopathic short stature. J Clin Endocrinol Metab. 2009 Feb;94(2):483-90. doi: 10.1210/jc.2008-1503. Epub 2008 Nov 11. PMID 19001519
- [Derived] Decker R, Albertsson-Wikland K, Kristrom B, Halldin M, Gustafsson J, Nilsson NO, Dahlgren J. GH Dose Reduction Maintains Normal Prepubertal Height Velocity After Initial Catch-Up Growth in Short Children. J Clin Endocrinol Metab. 2019 Mar 1;104(3):835-844. doi: 10.1210/jc.2018-01006. PMID 30339244
- Available data/document: Study Protocol — http://www.gpgrc.gu.se — The document will be found under "Trials" and then "GH-dose/Maintenance study"
- Available data/document: Statistical Analysis Plan — http://www.gpgrc.gu.se — The document will be found under "Trials" and then "GH-dose/Maintenance study"

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All children in the fix dose group and children in the individualized dose group who have reached their midparental height SDS (>- 0.6 SDS) during at least two years of GH-treatment within the 'GH-dose-catch up' study (TR 98-0198-003) and still are prepubertal were eligible in the study.
Pre-assignment Details: If glucose levels at the day of inclusion were higher than 7.1 mmol/L, then the child was excluded before assignment.
Groups:
- Decreased GH Dose: Decreased GH dose Genotropin
  Genotropin: Children were randomized to 50% GH dose after 2-3 years of initial GH treatment in previous trial (years depending on achieved Catch-up)
- Unchanged GH Dose: Unchanged GH dose
  Genotropin: Children were randomized to unchanged dose after 2-3 years of initial GH treatment in previous trial (years depending on achieved Catch-up)
- Control Group: Control Group with informed consent but not randomized
Period: Overall Study
Arm/Group | Decreased GH Dose | Unchanged GH Dose | Control Group
Started (observe that 33 more Children were included in the fix-arm (not randomized).) | 27 | 38 | 33
Completed | 23 | 32 | 31
Not Completed | 4 | 6 | 2

BASELINE CHARACTERISTICS:
Population: 98 children participated with two randomized arms (n=27+38) and one control arm with conventional fixed GH treatment (n=33).
Groups:
- Decreased GH Dose: Reduced dose 50% Genotropin
  Genotropin: Children were randomized to decreased GH dose by 50% after 2-3 years of Catch-up growth
- Unchanged GH Dose: Unchanged dose Genotropin
  Genotropin: Children were randomized to unchanged GH dose after 2-3 years of Catch-up growth
- Control Group: Control Group randomized in the previous study to fix dose.
  This group of children continued with fix dose in the current trial after signing informed consent.
- Total: Total of all reporting groups
Arm/Group | Decreased GH Dose | Unchanged GH Dose | Control Group | Total
Number analyzed (Participants) | 27 | 38 | 33 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 27 | 38 | 33 | 98
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.53 (1.51) | 8.52 (2.11) | 8.33 (1.78) | 8.52 (1.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 8 | 26
  Male | 20 | 27 | 25 | 72
Region of Enrollment [Number; unit: participants]
  Sweden | 27 | 38 | 33 | 65

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Children Maintaining Normal Growth Velocity
Description: The proportion of children in the intervention 1 group (=reduced dose) that maintained an individual ΔheightSDS within ±0.3 during the first year of the Maintenance trial, compared to the proportion of children in the intervention 2 group (non-reduced dose)
Time Frame: twelve months
Measure: Count of Participants; unit: Participants
Groups:
- Interventional 2: Unchanged GH dose
  Genotropin: Children were randomized to unchanged dose after 2-3 years of initial GH treatment in previous trial (years depending on achieved Catch-up)
- Control Group: Control Group children with fix dose through the previous and current trial and with signed consent
Arm/Group | Decreased GH Dose | Interventional 2 | Control Group
Number analyzed (Participants) | 27 | 38 | 33
Participants | 23 | 32 | 31

2. Secondary Outcome: IGF-I
Description: Delta Insulin-like growth factor-I (24 months after start compared to start of study) expressed as ng/ml and converted to standard deviation scores (SDS) to adjust for gender and age.
  A standard deviation score of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. A mean value within +-0.5 SDS and a range within +-1.0 SDS is a favorable outcome.
Time Frame: start of study to two years after start in the trial
Population: Drop outs due to puberty or adverse events
Measure: Mean (Standard Deviation); unit: standard deviation scores
Groups:
- Unchanged Dose: Unchanged dose Genotropin
  Genotropin: Children were randomized to unchanged GH dose after 2-3 years of Catch-up growth
- Reduced Dose: reduced dose 50% Genotropin
  Genotropin: Children were randomized to decreased GH dose by 50% after 2-3 years of Catch-up growth
- Control Group: Control Group treated with fix dose GH according to previous and current trial, with signed informed consent
Arm/Group | Unchanged Dose | Reduced Dose | Control Group
Number analyzed (Participants) | 15 | 22 | 23
standard deviation scores | -1.10 (1.14) | 0.58 (0.91) | -0.06 (1.26)

3. Secondary Outcome: Height SDS at Start of Puberty
Description: Height at start of puberty measured as cm and expressed as standard deviation score (SDS) to adjust for age and gender
Time Frame: 1-7 years in the trial
Population: All 98 Children were measured at start of puberty
Measure: Mean (Standard Deviation); unit: standard deviation scores
Groups:
- Decreased GH Dose: Children were randomized to decreased GH dose by 50% after 2-3 years of Catch-up growth
- Unchanged GH Dose: Children were randomized to unchanged GH dose after 2-3 years of Catch-up growth
- Control Group: Randomized in the previous study to fix dose. This Group of Children continued with fix dose in the current trial
Arm/Group | Decreased GH Dose | Unchanged GH Dose | Control Group
Number analyzed (Participants) | 27 | 38 | 33
standard deviation scores | -1.0 (1.02) | -1.06 (0.84) | -0.98 (0.91)

4. Other Pre Specified Outcome: Changes in Height
Description: Changes in height standard deviation scores (SDS) (calculated as height in cm at start converted to SDS and height in cm after two years in the trial converted to SDS)
Time Frame: start of study to two years after start in the trial
Measure: Mean (Standard Deviation); unit: standard deviation scores
Groups:
- Unchanged Dose: Unchanged dose Genotropin
  Genotropin: Children were randomized to either decreased dose by 50% or unchanged dose after 2-3 years of Catch-up growth
- Reduced Dose: reduced dose 50% Genotropin
  Genotropin: Children were randomized to either decreased dose by 50% or unchanged dose after 2-3 years of Catch-up growth
- Control Group: Control Group with fix dose throughout the previous and current trial. Signed informed consent.
Arm/Group | Unchanged Dose | Reduced Dose | Control Group
Number analyzed (Participants) | 15 | 22 | 23
standard deviation scores | 0.18 (0.16) | 0.57 (0.36) | 0.55 (0.26)

ADVERSE EVENTS:
Time Frame: Two years or in some cases up to seven prepubertal years
Description: No relevant information according to reviewer.
Groups:
- Decreased GH Dose: Reduced dose 50% Genotropin Children were randomized to decreased GH dose by 50% after 2-3 years of Catch-up growth
- Unchanged GH Dose: Unchanged dose
  Children were randomized to unchanged dose after 2-3 years of Catch-up growth
- Control Group: Control Group with fix dose.
  Children that were randomized to fix dose in the previous and current trial and signed informed consent
Arm/Group | Decreased GH Dose | Unchanged GH Dose | Control Group
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/38 | 0/33
Serious Adverse Events (participants affected / at risk) | 3/27 | 4/38 | 3/33
Other Adverse Events (participants affected / at risk) | 20/27 | 25/38 | 24/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decreased GH Dose (N=27) | Unchanged GH Dose (N=38) | Control Group (N=33)
Otitis media (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) — Otitis media with perforation needed hospitalization
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) — Hospitalization for risk of appendicitis
facial nerve palsy due to tick disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Hospitalization due to need for intravenous antibiotic treatment
accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Hospitalization due to car accident
fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) — Fracture after falling from a tree
Urinary tract infection (upper) (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) — Urinary tract infection with hospitalization
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decreased GH Dose (N=27) | Unchanged GH Dose (N=38) | Control Group (N=33)
virosis (Infections and infestations) | 20 (52) | 25 (46) | 24 (53) — Common adverse event was virosis winter-time

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No